CLINICAL TRIAL: NCT04924660
Title: CONNECTS Master Protocol for Clinical Trials Targeting Macro-, Micro-immuno-thrombosis, Vascular Hyperinflammation, and Hypercoagulability and Renin-angiotensin-aldosterone System (RAAS) in Hospitalized Patients With COVID-19 (ACTIV-4 Host Tissue)
Brief Title: Novel Experimental COVID-19 Therapies Affecting Host Response
Acronym: NECTAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sean Collins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Sean Collins, Professor, Emergency Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210982
Record Dates: First submitted 2021-06-09; First posted 2021-06-14 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; SARS-CoV-2 Infection; Coronavirus Infection
Keywords: COVID-19 drug treatment; RAAS
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — angiotensin I (1-7); Sar-Arg-Val-Tyr-Ile-His-Pro-Ala-OH; fostamatinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a two-step process: 1) The participant will first be randomized in an m:1 ratio to receive an active study drug or placebo, where m represents the number of study drug arms for which the participant is eligible. 2) The participant will then be randomly assigned with equal probability to one of the study drug arms. Participants will receive the corresponding study drug or matching placebo.
  Results data includes data from NCT05593770.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Which study drug arm the participant enters will be known to the research sites and the participants, but assignment to active versus placebo will be blinded. The randomized assignment, concealed from the research team, will be transmitted to the site pharmacy, who will provide study medication. The participant, treating clinicians, study personnel (other than the unblinded statistician who will prepare closed DSMB interim reports), and outcome assessors will all remain blinded to group assignment until after the database is locked and blinded analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TXA127 (4/20/2022 Arm Closed to Accrual) (Experimental): An investigational peptide agonist of Mas receptors.
  Interventions: Drug: TXA127
- TRV027 (4/20/2022 Arm Closed to Accrual) (Experimental): An investigational peptide biased agonist of the AT1 receptor.
  Interventions: Drug: TRV027
- Placebo (Placebo Comparator): NaCl 0.9% infused to match the duration of the agent for TXA127, TRV027, and APN01.
  Orange film-coated, plain, bioconvex tablets for fostamatinib.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
  Interventions: Drug: Placebo
- Fostamatinib (Experimental): An investigational oral spleen tyrosine kinase inhibitor.
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: TXA127 — TXA127 0.5 mg/kg/day infused 3 hours daily for 5 days or until hospital discharge whichever comes first.
  Arms: TXA127 (4/20/2022 Arm Closed to Accrual)
Drug: TRV027 — TRV027 12mg/h as a continuous 24-hour infusion, infused for 5 days or until hospital discharge whichever comes first.
  Arms: TRV027 (4/20/2022 Arm Closed to Accrual)
Drug: Placebo — NaCl 0.9% infused to match the duration of the agent (3 hours for TXA127 and continuous 24-hour infusion for TRV027, over 30 minutes for APN01.
  Orange film-coated, plain bioconvex tablets orally twice daily for 14 days or 28 doses for fostamatinib. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  Arms: Placebo
Drug: Fostamatinib — Fostamatinib100-150mg orally twice daily for 14 days or 28 doses. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  Arms: Fostamatinib

SUMMARY:
The overarching goal of the Master Protocol is to find effective strategies for inpatient management of patients with COVID-19. Therapeutic goals for patients hospitalized for COVID-19 include hastening recovery and preventing progression to critical illness, multiorgan failure, or death. Our objective is to determine whether modulating the host tissue response improves clinical outcomes among patients with COVID-19. The primary analysis will include data from NCT05593770.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which causes coronavirus disease 2019 (COVID-19), has resulted in a global pandemic. The clinical spectrum of COVID-19 infection is broad, encompassing asymptomatic infection, mild upper respiratory tract illness, and severe viral pneumonia with respiratory failure and death. Between 13 and 40% of patients become hospitalized, up to 30% of those hospitalized require admission for intensive care, and there is a 13% inpatient mortality rate. The reasons for hospitalization include respiratory support, as well as support for failure of other organs, including the heart and kidneys. The risk of thrombotic complications is increased, even when compared to other viral respiratory illnesses, such as influenza. While 82% of hospitalized patients with COVID-19 are ultimately discharged alive, median length of stay is 10-13 days.

Early work in treating COVID-19 has focused on preventing worsening of the initial clinical presentation to prevent hospitalization and disease progression to organ failure and death. Studies conducted under this Master Host Tissue Protocol are expected to extend our knowledge of how to manage patients who are hospitalized for COVID-19 illness. Our objective is to determine whether modulating the host tissue response improves clinical outcomes among patients with COVID-19. This Master Protocol is a randomized, placebo-controlled trial of agents targeting the host response in COVID-19 in hospitalized patients with hypoxemia. The Master Host Tissue Protocol is designed to be flexible in the number of study arms, the use of a single placebo group, and the stopping and adding of new therapies. Our primary outcome is oxygen free days through day 28. This is defined as days alive and without supplemental oxygen use during the first 28 days following randomization. Patients who die on or before day 28 are assigned -1 oxygen free days.

April 20, 2022 TRV027 and TXA127 arms closed to accrual.

ELIGIBILITY:
Inclusion criteria

1. Hospitalized for COVID-19
2. ≥18 years of age
3. SARS-CoV-2 infection, documented by:

   1. a nucleic acid test (NAT) or equivalent testing within 3 days prior to randomization OR
   2. documented by NAT or equivalent testing more than 3 days prior to randomization AND progressive disease suggestive of ongoing SARS-CoV-2 infection per the responsible investigator (For non-NAT tests, only those deemed with equivalent specificity to NAT by the protocol team will be allowed. A central list of allowed non- NAT tests is maintained in Appendix E. Appendix E. Non-NAT Tests Deemed with Equivalent Specificity to NAT by the Protocol Team).
4. Hypoxemia, defined as SpO2 <92% on room air, new receipt of supplemental oxygen to maintain SpO2 ≥92%, or increased supplemental oxygen to maintain SpO2 ≥92% for a patient on chronic oxygen therapy
5. Symptoms or signs of acute COVID-19, defined as one or more of the following:

   1. cough
   2. reported or documented body temperature of 100.4 degrees Fahrenheit or greater
   3. shortness of breath
   4. chest pain
   5. infiltrates on chest imaging (x-ray, CT scan, lung ultrasound)

Exclusion criteria

1. Onset of COVID-19 symptom fulfilling inclusion criterion #5 >14 days prior to randomization
2. Hospitalized with hypoxemia (as defined in inclusion #4) for >72 hours prior to randomization (the 72-hour window for randomization begins when the patient first meets the hypoxemia inclusion criteria after hospital admission)
3. Pregnancy
4. Breastfeeding
5. Prisoners
6. End-stage renal disease (ESRD) on dialysis
7. Patient undergoing comfort care measures only such that treatment focuses on end-of-life symptom management over prolongation of life.
8. The treating clinician expects inability to participate in study procedures or participation would not be in the best interests of the patient
9. Known allergy/hypersensitivity to IMP or its excipients

The following exclusion criteria differ from the master protocol criteria:

TXA127-specific exclusion criteria(4/20/2022 Closed to Accrual):

1. Patient unable to participate or declines participation in the TXA127/Ang(1-7) arm.
2. History of sensitivity (including angioedema) or allergic reaction to medication targeting the RAAS system including study medications or other allergy in the opinion of the investigator that contraindicates participation (not applicable to fostamatinib arm)
3. Hemodynamic instability - defined as MAP < 65 mmHg at time of randomization confirmed on two measurements 5 minutes apart OR vasopressors at or above norepinephrine equivalent of 0.1 mcg/kg/min in prior 4 hours to maintain MAP > 65 mmHg.
4. Known severe renal artery stenosis.
5. Known significant left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic or mitral stenosis.
6. Randomized in another trial evaluating RAAS modulation in the prior 30 days

TRV027-specific exclusion criteria (4/20/2022 Closed to Accrual):

1. Participants on ARBs will be excluded from this study arm.
2. Patient unable to participate or declines participation in the TRV027 arm.
3. History of sensitivity (including angioedema) or allergic reaction to medication targeting the RAAS system including study medications or other allergy in the opinion of the investigator that contraindicates participation (not applicable to fostamatinib arm)
4. Hemodynamic instability - defined as MAP < 65 mmHg at time of randomization confirmed on two measurements 5 minutes apart OR vasopressors at or above norepinephrine equivalent of 0.1 mcg/kg/min in prior 4 hours to maintain MAP > 65 mmHg.
5. Known severe renal artery stenosis.
6. Known significant left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic or mitral stenosis.
7. Randomized in another trial evaluating RAAS modulation in the prior 30 days

Fostamatinib specific exclusion criteria:

The following exclusion criteria differ from the master protocol criteria:

1. Randomized in another trial evaluating fostamatinib in the prior 30 days

Study arm exclusion criteria measured within 24 hours prior to randomization:

1. AST or ALT ≥ 5 × upper limit of normal (ULN) or ALT or AST ≥ 3 × ULN and total bilirubin ≥ 2 × ULN
2. SBP > 160 mmHg or DBP > 100 mmHg at the time of screening and randomization
3. ANC < 1000/mL
4. Patient is anticipated to require a strong CYP3A inhibitor (Atazanavir, Certinib, Clarithromycin, Cobicistat and cobicistat-containing coformulations, Idelalisib,Indinavir, Itraconazole, Ketoconazole, Levoketoconazole, Lonafarnib, Lopinavir, Mifeprostone, Mibefradil, Nefazodone, Nelfinavir, Ombitasvir-paritaprevir-ritonavir plus dasabuvir, Posaconazole, Ribociclib Ritonavir, Saquinavir, Telithromycin, Troleandomycin, Tucatinib, Voriconazole) from randomization to 21 days post-randomization. For a full list of CYP3A4 substrates, please reference this regularly updated list: https://drug-interactions.medicine.iu.edu/MainTable.aspx.
5. Patient unable to participate or declines participation in the fostamatinib arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. Collins, M.D., Study Chair — Vanderbilt University Medical Center
Locations (51):
- United States (51):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Public Health Trust of Miami-Dade County, Florida - Jackson Memorial Hospital, Miami, Florida
  - Ponce de Leon Clinical Research Site, Atlanta, Georgia
  - Emory Johns Creek, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - AMITA Health St. Alexius Medical Center, Hoffman Estates, Illinois
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center Weiler Campus, The Bronx, New York
  - Montefiore Medical Center Moses Campus, The Bronx, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - West Chester Hospital, West Chester, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - UVA Health, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Health, Richmond, Virginia
  - Harborview Medical Center/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collins SP, Shotwell MS, Strich JR, Gibbs KW, de Wit M, Files DC, Harkins M, Hudock K, Merck LH, Moskowitz A, Apodaca KD, Barksdale A, Safdar B, Javaheri A, Sturek JM, Schrager H, Iovine NM, Tiffany B, Douglas I, Levitt J, Ginde AA, Hager DN, Shapiro N, Duggal A, Khan A, Lanspa M, Chen P, Gentile N, Harris E, Gong M, Sellers S, Goodwin AJ, Tidswell MA, Filbin M, Desai N, Gutierrez F, Estrada V, Burgos J, Boyles T, Pano-Pardo JR, Hussen N, Rosenberg Y, Troendle J, Bernard GR, Bistran-Hall AJ, Walsh K, Casey JD, DeClercq J, Joly MM, Pulley J, Rice TW, Schildcrout JS, Wang L, Semler MW, Self WH; ACTIV-4 Host Tissue Investigators. Fostamatinib for Hospitalized Adults With COVID-19 and Hypoxemia: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2448215. doi: 10.1001/jamanetworkopen.2024.48215. PMID 39625722
- [Derived] Self WH, Shotwell MS, Gibbs KW, de Wit M, Files DC, Harkins M, Hudock KM, Merck LH, Moskowitz A, Apodaca KD, Barksdale A, Safdar B, Javaheri A, Sturek JM, Schrager H, Iovine N, Tiffany B, Douglas IS, Levitt J, Busse LW, Ginde AA, Brown SM, Hager DN, Boyle K, Duggal A, Khan A, Lanspa M, Chen P, Puskarich M, Vonderhaar D, Venkateshaiah L, Gentile N, Rosenberg Y, Troendle J, Bistran-Hall AJ, DeClercq J, Lavieri R, Joly MM, Orr M, Pulley J, Rice TW, Schildcrout JS, Semler MW, Wang L, Bernard GR, Collins SP; ACTIV-4 Host Tissue Investigators. Renin-Angiotensin System Modulation With Synthetic Angiotensin (1-7) and Angiotensin II Type 1 Receptor-Biased Ligand in Adults With COVID-19: Two Randomized Clinical Trials. JAMA. 2023 Apr 11;329(14):1170-1182. doi: 10.1001/jama.2023.3546. PMID 37039791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This adaptive platform study consisted of 3 trials, each designed to assess a candidate agent as treatment for coronavirus disease 2019 (COVID-19) in hospitalized adult patients who had severe infection with acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes COVID-19. The control group for each trial includes all participants that were eligible for that trial and received a placebo mimic for any of the three study agents (shared placebo).
Pre-assignment Details: Adults hospitalized with COVID-19 were enrolled with no exclusions based on age, sex, race, ethnicity, severity of disease or preferred language. If a patient appeared to meet eligibility criteria, the site investigator approached the treating clinician to ask permission to approach the patient to confirm eligibility, discuss potential study recruitment, and proceed with informed consent. The eligibility criteria were verified and informed consent was obtained just prior to randomization.
Groups:
- TXA127 Shared Placebo: NaCl 0.9% infused to match the duration (3 hours) of the agent for TXA127. (3 hours for TXA127
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
- TRV027 Shared Placebo: NaCl 0.9% infused to match the duration(continuous 24-hour infusion) of the agent for TRV027.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
- Fostamatinib Shared Placebo: Orange film-coated, plain biconvex tablets orally twice daily for 14 days or 28 doses for fostamatinib placebo. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
Period: United States
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 176 | 175 | 149 | 147 | 193 | 192
Completed | 124 | 130 | 99 | 114 | 140 | 145
Not Completed | 52 | 45 | 50 | 33 | 53 | 47
Not completed — Death | 29 | 32 | 34 | 25 | 26 | 23
Not completed — Lost to Follow-up | 15 | 10 | 13 | 5 | 19 | 20
Not completed — Withdrawal by Subject | 8 | 3 | 3 | 3 | 8 | 4
Period: Spain
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 0 | 0 | 0 | 0 | 10 | 9
Completed | 0 | 0 | 0 | 0 | 9 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Brazil
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 0 | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Period: Germany
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 0 | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Italy
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 0 | 0 | 0 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: South Africa
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Started | 0 | 0 | 0 | 0 | 2 | 3
Completed | 0 | 0 | 0 | 0 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo | Total
Number analyzed (Participants) | 176 | 175 | 149 | 147 | 207 | 206 | 1060
Age, Categorical [Count of Participants; unit: Participants] — Population: Results data includes data from NCT05593770. All Countries = all participant data The remaining rows are data by country.
  Participants
    All Countries: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    All Countries: Between 18 and 65 years | 121 | 128 | 109 | 107 | 88 | 81 | 634
    All Countries: >=65 years | 55 | 47 | 40 | 40 | 119 | 125 | 426
    United States: number analyzed (Participants) | 176 | 175 | 149 | 147 | 193 | 192 | 1032
    United States: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    United States: Between 18 and 65 years | 121 | 128 | 109 | 107 | 84 | 78 | 627
    United States: >=65 years | 55 | 47 | 40 | 40 | 109 | 114 | 405
    Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 19
    Spain: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: Between 18 and 65 years | 0 | 0 | 0 | 0 | 2 | 2 | 4
    Spain: >=65 years | 0 | 0 | 0 | 0 | 8 | 7 | 15
    Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: Between 18 and 65 years | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: >=65 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Italy: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: >=65 years | 0 | 0 | 0 | 0 | 1 | 1 | 2
    South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 5
    South Africa: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Between 18 and 65 years | 0 | 0 | 0 | 0 | 1 | 1 | 2
    South Africa: >=65 years | 0 | 0 | 0 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Results data includes data from NCT05593770. All Countries = all participant data The remaining rows are data by country.
  Participants
    All Countries: Female | 70 | 76 | 54 | 69 | 103 | 95 | 467
    All Countries: Male | 106 | 99 | 95 | 78 | 104 | 111 | 593
    United States: number analyzed (Participants) | 176 | 175 | 149 | 147 | 193 | 192 | 1032
    United States: Female | 70 | 76 | 54 | 69 | 97 | 89 | 455
    United States: Male | 106 | 99 | 95 | 78 | 96 | 103 | 577
    Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 19
    Spain: Female | 0 | 0 | 0 | 0 | 3 | 4 | 7
    Spain: Male | 0 | 0 | 0 | 0 | 7 | 5 | 12
    Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: Female | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Male | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Italy: Female | 0 | 0 |  |  | 1 | 1 | 2
    Italy: Male | 0 | 0 |  |  | 0 | 0 | 0
    South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 5
    South Africa: Female | 0 | 0 | 0 | 0 | 1 | 1 | 2
    South Africa: Male | 0 | 0 | 0 | 0 | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Results data includes data from NCT05593770. All Countries = all participant data The remaining rows are data by country.
  Participants
    All Countries: Hispanic or Latino | 28 | 26 | 25 | 23 | 27 | 30 | 159
    All Countries: Not Hispanic or Latino | 140 | 140 | 113 | 116 | 174 | 165 | 848
    All Countries: Unknown or Not Reported | 8 | 9 | 11 | 8 | 6 | 11 | 53
    United States: number analyzed (Participants) | 176 | 175 | 149 | 147 | 193 | 192 | 1032
    United States: Hispanic or Latino | 28 | 26 | 25 | 23 | 21 | 25 | 148
    United States: Not Hispanic or Latino | 140 | 140 | 113 | 116 | 170 | 161 | 840
    United States: Unknown or Not Reported | 8 | 9 | 11 | 8 | 2 | 6 | 44
    Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 19
    Spain: Hispanic or Latino | 0 | 0 | 0 | 0 | 5 | 5 | 10
    Spain: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Spain: Unknown or Not Reported | 0 | 0 | 0 | 0 | 4 | 4 | 8
    Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: Hispanic or Latino |  |  |  | 0 | 0 | 0 | 0
    Brazil: Not Hispanic or Latino |  |  |  | 0 | 0 | 0 | 0
    Brazil: Unknown or Not Reported |  |  |  | 0 | 1 | 0 | 1
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Italy: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Italy: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
    South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 5
    South Africa: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Not Hispanic or Latino | 00 | 0 | 0 | 0 | 2 | 3 | 5
    South Africa: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Results data includes data from NCT05593770. All Countries = all participant data The remaining rows are data by country.
  Participants
    All Countries: American Indian or Alaska Native | 5 | 1 | 2 | 1 | 2 | 4 | 15
    All Countries: Asian | 4 | 4 | 2 | 3 | 6 | 6 | 25
    All Countries: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 3 | 0 | 4
    All Countries: Black or African American | 29 | 30 | 25 | 22 | 24 | 23 | 153
    All Countries: White | 115 | 114 | 101 | 97 | 149 | 160 | 736
    All Countries: More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 2
    All Countries: Unknown or Not Reported | 22 | 25 | 19 | 24 | 22 | 13 | 125
    United States: number analyzed (Participants) | 176 | 175 | 149 | 147 | 193 | 192 | 1032
    United States: American Indian or Alaska Native | 5 | 1 | 2 | 1 | 2 | 4 | 15
    United States: Asian | 4 | 4 | 2 | 3 | 6 | 6 | 25
    United States: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 3 | 0 | 4
    United States: Black or African American | 29 | 30 | 25 | 22 | 22 | 21 | 149
    United States: White | 115 | 114 | 101 | 97 | 139 | 148 | 714
    United States: More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 2
    United States: Unknown or Not Reported | 22 | 25 | 19 | 24 | 20 | 13 | 123
    Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9 | 19
    Spain: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: White | 0 | 0 | 0 | 0 | 9 | 9 | 18
    Spain: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Spain: Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Brazil: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: White | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Brazil: Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: White | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Germany: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Germany: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Italy: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: White | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Italy: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Italy: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 5
    South Africa: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Black or African American | 0 | 0 | 0 | 0 | 2 | 2 | 4
    South Africa: White | 0 | 0 | 0 | 0 | 0 | 1 | 1
    South Africa: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    South Africa: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 176 | 175 | 149 | 147 | 193 | 192 | 871
  Spain | 0 | 0 | 0 | 0 | 10 | 9 | 19
  Brazil | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Italy | 0 | 0 | 0 | 0 | 1 | 1 | 2
  South Africa | 0 | 0 | 0 | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Free Days Through Day 28.
Description: This is defined as days alive and without supplemental oxygen use during the first 28 days following randomization. Patients who die on or before day 28 are assigned -1 oxygen free days. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO).
Time Frame: Day 1 to Day 28
Population: Results data includes data from NCT05593770. All countries = all participant data. The 'Overall Number of Participants Analyzed' includes those with recorded outcomes, excluding ineligible participants or those who didn't receive the treatment. It reflects contributors to CT.gov outcome summaries. Some outcomes before day 90 may inflate this number. Participants who lacked outcome data were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- TXA127 Placebo: NaCl 0.9% infused to match the duration (3 hours) of the agent for TXA127. (3 hours for TXA127
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
- TRV027 Placebo: NaCl 0.9% infused to match the duration(continuous 24-hour infusion) of the agent for TRV027.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
- Fostamatinib Placebo: Orange film-coated, plain biconvex tablets orally twice daily for 14 days or 28 doses for fostamatinib placebo. Study medication will be continued as an outpatient if the patient is discharged prior to completing 28 doses.
  For the purposes of interim and final analyses, the route and frequency of placebo will be ignored, and all placebo participants will be pooled together as a single group. In comparing an active drug versus placebo, only those placebo participants that were eligible for the active drug will be included.
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Placebo | Fostamatinib | Fostamatinib Placebo
Number analyzed (Participants) | 153 | 155 | 135 | 131 | 177 | 181
Days
  All Countries | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 13.4 (12.4) | 14.2 (12.1)
  United States: number analyzed (Participants) | 153 | 155 | 135 | 131 | 164 | 170
  United States | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 12.9 (12.5) | 13.9 (12)
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 8
  Spain |  |  |  |  | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil |  |  |  |  | -1 (NA) — Unable to provide standard deviation only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany |  |  |  |  |  | 0 (NA) — Unable to provide standard deviation only 1 participant affected
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy |  |  |  |  | 14 (NA) — Unable to provide standard deviation only 1 participant affected |
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa |  |  |  |  | 25.5 (3.5) | 26.5 (0.7)

2. Secondary Outcome: In-hospital Mortality
Description: Number of patients who die during hospitalization
Time Frame: Day 1 to hospital discharge or Day 90 whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 167 | 172 | 145 | 144 | 197 | 197
Participants
  All Countries | 23 | 24 | 31 | 20 | 23 | 16
  United States: number analyzed (Participants) | 167 | 172 | 145 | 144 | 184 | 185
  United States | 23 | 24 | 31 | 20 | 22 | 15
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 1
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 1 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Alive and Oxygen Free at Day 14
Description: Number of patients oxygen free at day 14. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO).
Time Frame: Day 1 to Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 158 | 164 | 138 | 137 | 189 | 191
Participants
  All Countries | 60 | 86 | 48 | 66 | 113 | 113
  United States: number analyzed (Participants) | 158 | 164 | 138 | 137 | 176 | 179
  United States | 60 | 86 | 48 | 66 | 103 | 105
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 8 | 6
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 2 | 2
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Alive and Oxygen Free at Day 28
Description: Number of patients oxygen-free at day 28. Patients will be considered to be receiving supplemental oxygen therapy when they are receiving any of the following: supplemental oxygen by nasal cannula, supplemental oxygen by face mask, high flow nasal cannula (HFNC), non-invasive ventilation (NIV), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO).
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 155 | 158 | 135 | 134 | 187 | 189
Participants
  All Countries | 78 | 87 | 60 | 69 | 106 | 123
  United States: number analyzed (Participants) | 155 | 158 | 135 | 134 | 174 | 177
  United States | 78 | 87 | 60 | 69 | 95 | 114
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 8 | 7
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 0 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 1 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 2 | 2

5. Secondary Outcome: Alive and Free of New Invasive Mechanical Ventilation at Day 28
Description: Number of patients alive free of new invasive mechanical ventilation at day 28
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 155 | 160 | 136 | 136 | 186 | 190
Participants
  All Countries | 124 | 128 | 99 | 109 | 160 | 171
  United States: number analyzed (Participants) | 155 | 160 | 136 | 136 | 173 | 178
  United States | 124 | 128 | 99 | 109 | 148 | 160
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 9 | 8
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 0 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 1
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 1 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 2 | 2

6. Secondary Outcome: 28-day Mortality
Description: Number of patients who have died at Day 28
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 163 | 166 | 141 | 140 | 195 | 197
Participants
  All Countries | 22 | 22 | 29 | 18 | 22 | 16
  United States: number analyzed (Participants) | 163 | 166 | 141 | 140 | 182 | 185
  United States | 22 | 22 | 29 | 18 | 21 | 15
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 1
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 1 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: 60-day Mortality
Description: Number of patients who have died at Day 60
Time Frame: Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 161 | 166 | 139 | 140 | 195 | 195
Participants
  All Countries | 26 | 29 | 33 | 23 | 25 | 22
  United States: number analyzed (Participants) | 161 | 166 | 139 | 140 | 182 | 183
  United States | 26 | 29 | 33 | 23 | 24 | 20
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 2
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 1 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: 90-day Mortality
Description: Number of patients who have died at Day 90
Time Frame: Day 90
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 158 | 161 | 135 | 138 | 186 | 186
Participants
  All Countries | 28 | 31 | 34 | 25 | 27 | 26
  United States: number analyzed (Participants) | 158 | 161 | 135 | 138 | 174 | 174
  United States | 28 | 31 | 34 | 25 | 26 | 23
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 2
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 1 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa | 0 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Clinical Status Assessed Using World Health Organization(WHO) 8-point Ordinal Scale
Description: Number of participants who fell within the ordinal scale per the below criteria. Each row represents the country and number of participants with the score in numerical order.
  1. Ambulatory - Not hospitalized and no limitation of activities
  2. Ambulatory - Not hospitalized with limitation of activities or home oxygen use
  3. Hospitalized Mild Disease - Hospitalized, no oxygen therapy
  4. Hospitalized Mild Disease - Hospitalized, oxygen by mask or nasal prongs
  5. Hospitalized Severe Disease - Non-invasive ventilation or high-flow nasal cannula
  6. Hospitalized Severe Disease -Invasive mechanical ventilation
  7. Hospitalized Severe Disease - Invasive mechanical ventilation plus additional organ support with- vasopressors, RRT, or ECMO
  8. Dead
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 158 | 164 | 138 | 137 | 188 | 191
Participants
  Alll Countries Score=1 | 37 | 57 | 31 | 45 | 53 | 75
  Alll Countries Score=2 | 61 | 53 | 50 | 48 | 79 | 77
  Alll Countries Score=3 | 5 | 5 | 2 | 3 | 15 | 4
  Alll Countries Score=4 | 19 | 7 | 8 | 6 | 20 | 14
  Alll Countries Score=5 | 6 | 7 | 7 | 6 | 3 | 2
  Alll Countries Score=6 | 6 | 6 | 5 | 4 | 4 | 2
  Alll Countries Score =7 | 12 | 14 | 14 | 14 | 3 | 7
  Alll Countries Score=8 | 12 | 13 | 21 | 11 | 11 | 10
  United States Score=1: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=1 | 37 | 57 | 31 | 45 | 45 | 68
  United States Score=2: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=2 | 61 | 55 | 50 | 48 | 76 | 59
  United States Score=3: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=3 | 5 | 5 | 2 | 3 | 15 | 3
  United States Score=4: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=4 | 19 | 7 | 8 | 6 | 19 | 11
  United States Score=5: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=5 | 6 | 7 | 7 | 6 | 3 | 2
  United States Score=6: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=6 | 6 | 6 | 8 | 4 | 4 | 2
  United States Score=7: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=7 | 12 | 14 | 14 | 14 | 1 | 7
  United States Score=8: number analyzed (Participants) | 158 | 164 | 138 | 137 | 175 | 179
  United States Score=8 | 12 | 13 | 21 | 11 | 10 | 9
  Spain Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=1 | 0 | 0 | 0 | 0 | 6 | 5
  Spain Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=2 | 0 | 0 | 0 | 0 | 3 | 1
  Spain Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=4 | 0 | 0 | 0 | 0 | 0 | 2
  Spain Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=8 | 0 | 0 | 0 | 0 | 0 | 1
  Brazil Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=8 | 0 | 0 | 0 | 0 | 1 | 0
  Germany Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=4 | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=8 | 0 | 0 | 0 | 0 | 0 | 0
  Italy=Score1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy=Score1 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=4 | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=8 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=1 | 0 | 0 | 0 | 0 | 2 | 1
  South Africa Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=3 | 0 | 0 | 0 | 0 | 0 | 1
  South Africa Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=8 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Clinical Status Assessed Using WHO 8-point Ordinal Scale at Day 28
Description: as for outcome 9
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 154 | 158 | 135 | 134 | 182 | 189
Participants
  All Countries Score=1 | 58 | 62 | 48 | 47 | 63 | 74
  All Countries Score=2 | 53 | 58 | 44 | 53 | 76 | 88
  All Countries Score=3 | 4 | 2 | 0 | 2 | 6 | 3
  All Countries Score=4 | 7 | 1 | 3 | 2 | 8 | 3
  All Countries Score=5 | 1 | 3 | 3 | 3 | 1 | 2
  All Countries Score=6 | 4 | 5 | 3 | 4 | 1 | 1
  All Countries Score=7 | 5 | 5 | 5 | 5 | 3 | 2
  All Countries Score=8 | 22 | 22 | 29 | 18 | 22 | 16
  United States Score=1: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=1 | 58 | 62 | 48 | 47 | 56 | 67
  United States Score=2: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=2 | 53 | 58 | 44 | 53 | 75 | 85
  United States Score=3: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=3 | 4 | 2 | 0 | 2 | 5 | 2
  United States Score=4: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=4 | 7 | 2 | 3 | 2 | 7 | 3
  United States Score=5: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=5 | 1 | 3 | 3 | 3 | 1 | 2
  United States Score=6: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=6 | 4 | 5 | 3 | 4 | 1 | 1
  United States Score=7: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=7 | 5 | 5 | 5 | 5 | 3 | 2
  United States Score=8: number analyzed (Participants) | 154 | 158 | 135 | 134 | 169 | 177
  United States Score=8 | 22 | 22 | 29 | 18 | 21 | 15
  Spain Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=1 | 0 | 0 | 0 | 0 | 7 | 6
  Spain Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=2 | 0 | 0 | 0 | 0 | 0 | 2
  Spain Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=3 | 0 | 0 | 0 | 0 | 1 | 0
  Spain Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=4 | 0 | 0 | 0 | 0 | 1 | 0
  Spain Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain Score=8 | 0 | 0 | 0 | 0 | 0 | 1
  Brazil Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=8 | 0 | 0 | 0 | 0 | 1 | 0
  Germany Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=2 | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=8 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=2 | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Italy Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy Score=8 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=1 | 0 | 0 | 0 | 0 | 2 | 1
  South Africa Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=3 | 0 | 0 | 0 | 0 | 0 | 1
  South Africa Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=8 | 0 | 0 | 0 | 0 | 0 | 1

11. Secondary Outcome: Clinical Status Assessed Using WHO 8-point Ordinal Scale at Day 60
Description: as for outcome 9
Time Frame: Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 128 | 140 | 108 | 115 | 161 | 167
Participants
  All Countries Score=1 | 37 | 57 | 31 | 45 | 53 | 75
  All Countries Score=2 | 61 | 55 | 50 | 48 | 79 | 77
  All Countries Score=3 | 5 | 5 | 2 | 3 | 15 | 4
  All Countries Score=4 | 19 | 7 | 8 | 6 | 20 | 14
  All Countries Score=5 | 6 | 7 | 7 | 6 | 3 | 2
  All Countries Score=6 | 6 | 9 | 5 | 4 | 4 | 2
  All Countries Score=7 | 12 | 14 | 14 | 14 | 3 | 7
  All Countries Score=8 | 12 | 13 | 21 | 21 | 11 | 10
  United States Score=1: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=1 | 37 | 57 | 31 | 45 | 45 | 69
  United States Score=2: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=2 | 61 | 55 | 50 | 48 | 76 | 76
  United States Score=3: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=3 | 5 | 5 | 2 | 3 | 15 | 3
  United States Score=4: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=4 | 19 | 7 | 8 | 6 | 19 | 11
  United States Score=5: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=5 | 6 | 7 | 7 | 6 | 3 | 2
  United States Score=6: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=6 | 6 | 6 | 5 | 4 | 4 | 2
  United States Score=7: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=7 | 12 | 14 | 14 | 14 | 3 | 7
  United States Score=8: number analyzed (Participants) | 128 | 140 | 108 | 115 | 150 | 155
  United States Score=8 | 12 | 13 | 21 | 11 | 10 | 9
  Spain Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=1 | 0 | 0 | 0 | 0 | 5 | 6
  Spain Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=2 | 0 | 0 | 0 | 0 | 2 | 1
  Spain Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=4 | 0 | 0 | 0 | 0 | 1 | 0
  Spain Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Spain Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  Spain Score=8 | 0 | 0 | 0 | 0 | 0 | 2
  Brazil Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Brazil Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil Score=8 | 0 | 0 | 0 | 0 | 1 | 0
  Germany Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=1 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=3 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=4 | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  Germany Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany Score=8 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=1 | 0 | 0 | 0 | 0 | 2 | 1
  South Africa Score=2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=2 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=3 | 0 | 0 | 0 | 0 | 0 | 1
  South Africa Score=4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=4 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=5 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=6 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=7 | 0 | 0 | 0 | 0 | 0 | 0
  South Africa Score=8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa Score=8 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Hospital-free Days Through Day 28
Description: Days alive and not hospitalized during the first 28 days following randomization. Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 154 | 160 | 136 | 136 | 184 | 190
Days
  All Countries | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 13.4 (12.4) | 14.2 (12.1)
  United States: number analyzed (Participants) | 154 | 160 | 136 | 136 | 171 | 178
  United States | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 12.9 (12.5) | 13.9 (12)
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain |  |  |  |  | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil |  |  |  |  | -1 (NA) — Unable to provide standard deviation only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany |  |  |  |  |  | 0 (NA) — Unable to provide standard deviation only 1 participant affected
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy |  |  |  |  | 14 (NA) — Unable to provide standard deviation only 1 participant affected |
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa |  |  |  |  | 25.5 (3.5) | 26.5 (0.7)

13. Secondary Outcome: Ventilator-free Days Through Day 28
Description: Days alive and not receiving mechanical ventilation during the first 28 days following randomization. Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 150 | 159 | 135 | 135 | 177 | 186
Days
  All Countries | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 12.9 (12.5) | 13.9 (12)
  United States: number analyzed (Participants) | 150 | 159 | 135 | 135 | 164 | 174
  United States | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 12.9 (12.5) | 13.9 (12)
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain |  |  |  |  | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil |  |  |  |  | -1 (NA) — Unable to provide standard deviation only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany |  |  |  |  |  | 0 (NA) — Unable to provide standard deviation only 1 participant affected
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy |  |  |  |  | 14 (NA) — Unable to provide standard deviation only 1 participant affected |
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa |  |  |  |  | 25.5 (3.5) | 26.5 (0.7)

14. Secondary Outcome: Respiratory Failure-free Days Through Day 28
Description: Days alive and not in respiratory failure during the first 28 days following randomization. A respiratory failure-free day is defined as a day alive without the use of HFNC, NIV, IMV, or (ECMO). Patients who die on or before day 28 are assigned a value -1.
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 150 | 160 | 135 | 136 | 177 | 186
Days
  All Countries | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 13.4 (12.4) | 14.2 (12.1)
  United States: number analyzed (Participants) | 150 | 160 | 135 | 136 | 164 | 174
  United States | 9.0 (10.9) | 11.3 (11.5) | 8.1 (10.8) | 10.5 (11.5) | 12.9 (12.5) | 13.9 (12)
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain |  |  |  |  | 21.3 (8.2) | 19.5 (12.5)
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 177 | 0
  Brazil |  |  |  |  | -1 (NA) — Unable to provide standard deviation only 1 participant affected |
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany |  |  |  |  |  | 0 (NA) — Unable to provide standard deviation only 1 participant affected
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy |  |  |  |  | 14 (NA) — Unable to provide standard deviation only 1 participant affected |
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2
  South Africa |  |  |  |  | 25.3 (3.5) | 26.5 (0.7)

15. Other Pre Specified Outcome: Hypotension
Description: Number of participants with hypotension defined by low arterial blood pressure leading to either [1] initiation or increase in vasopressor therapy, [2] administration of a fluid bolus of 500 ml or more, or [3] modification of the dose or discontinuation of the study drug.
Time Frame: Day 0 to Day 5 or hospital discharge whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 170 | 173 | 145 | 145 | 199 | 201
Participants
  All Countries | 31 | 31 | 32 | 25 | 24 | 18
  United States: number analyzed (Participants) | 170 | 173 | 145 | 145 | 186 | 188
  United States | 31 | 31 | 32 | 25 | 23 | 17
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 1
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 1 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 1
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Allergic Reaction
Description: Number of participants with allergic reaction, including rash and angioedema
Time Frame: Day 0 to Day 5 or hospital discharge whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 170 | 173 | 145 | 145 | 199 | 201
Participants
  All Countries | 3 | 4 | 0 | 3 | 3 | 1
  United States: number analyzed (Participants) | 170 | 173 | 145 | 145 | 186 | 188
  United States | 3 | 4 | 0 | 3 | 3 | 1
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 0
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 0 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: Incident Renal Replacement Therapy During Hospitalization
Description: Number of participants requiring renal replacement therapy during hospitalization (when possible, at participating sites)
Time Frame: Day 0 to Day 5 or hospital discharge whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Shared Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Shared Placebo | Fostamatinib | Fostamatinib Shared Placebo
Number analyzed (Participants) | 170 | 173 | 145 | 145 | 199 | 201
Participants
  All Countries | 11 | 12 | 9 | 11 | 5 | 9
  United States: number analyzed (Participants) | 170 | 173 | 145 | 145 | 186 | 188
  United States | 11 | 12 | 9 | 11 | 15 | 9
  Spain: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  Spain | 0 | 0 | 0 | 0 | 0 | 0
  Brazil: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Brazil | 0 | 0 | 0 | 0 | 0 | 0
  Germany: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 0 | 0 | 0
  Italy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Italy | 0 | 0 | 0 | 0 | 0 | 0
  South Africa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3
  South Africa | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Serious and Non-Serious AEs include data for all countries. Results data includes data from NCT05593770.
Arm/Group | TXA127 (4/20/2022 Arm Closed to Accrual) | TXA127 Placebo | TRV027 (4/20/2022 Arm Closed to Accrual) | TRV027 Placebo | Fostamatinib | Fostamatinib Placebo
All-Cause Mortality (participants affected / at risk) | 29/176 | 32/175 | 34/149 | 25/147 | 27/193 | 26/192
Serious Adverse Events (participants affected / at risk) | 8/176 | 4/175 | 6/149 | 2/147 | 16/193 | 44/192
Other Adverse Events (participants affected / at risk) | 29/176 | 5/175 | 3/149 | 6/147 | 18/193 | 25/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA127 (4/20/2022 Arm Closed to Accrual) (N=176) | TXA127 Placebo (N=175) | TRV027 (4/20/2022 Arm Closed to Accrual) (N=149) | TRV027 Placebo (N=147) | Fostamatinib (N=193) | Fostamatinib Placebo (N=192)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection bacteria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulval cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA127 (4/20/2022 Arm Closed to Accrual) (N=176) | TXA127 Placebo (N=175) | TRV027 (4/20/2022 Arm Closed to Accrual) (N=149) | TRV027 Placebo (N=147) | Fostamatinib (N=193) | Fostamatinib Placebo (N=192)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oral Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT04924660/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT04924660/SAP_003.pdf
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04924660/ICF_001.pdf